CLINICAL TRIAL: NCT03280888
Title: Relevance of Peripheral Cells in the Pathophysiology of Chronic Myelomonocytic Leukemia (CMML)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 13-PP-11
Record Dates: First submitted 2017-01-31; First posted 2017-09-13 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Myelomonocytic Leukemia (CMML) is the most frequent of myelodysplastic/myeloproliferative syndromes, as defined by the WHO classification of myeloid malignancies. The median age at diagnosis is around 70 years with a strong male predominance. CMML is a clonal disease of the bone marrow hematopoietic stem cell mainly characterized by persistent monocytosis (>1x109/L) and the presence of immature dysplastic granulocytes in the peripheral blood of CMML patients. Allogeneic stem cell transplantation (ASCT) remains the only curative option in CMML. However, CMML patients are rarely eligible for this kind of therapy, mainly due to their advanced age. The gold standard treatment of CMML thus remains hydroxyurea, which is usually initiated when the disease becomes proliferative, and demethylating agents, which could be efficient in the most aggressive forms of CMML. Nevertheless, the pathogenesis of CMML remains poorly understood and new therapies are urgently needed for patients in treatment failure.

In recent years, a large numbers of gene mutations have been discovered in CMML, none of which are specific of this entity, as they can be encountered with different frequencies in other myeloid neoplasms. These mutated genes encode signaling molecules (NRAS, KRAS, CBL, JAK2, FLT3 and several members of the Notch pathway), epigenetic regulators (TET2, ASXL1, EZH2, IDH1, IDH2,.) and splicing factors (SF3B1, SRSF2, ZRSF2). Mutations in the transcription regulators RUNX1, NPM1 and TP53 have also been reported in CMML. However, the role of these mutations in leukemogenesis is still unclear. CMML is also characterized by defects in monocyte to macrophage differentiation. These defects in monocyte differentiation can be attributed to the presence of immature dysplastic granulocytes that secrete high levels of alpha-defensins HNP1-3 that antagonize the purinergic receptor P2RY6 in CMML patients. These CD14-/CD15+/CD24+ immature granulocytes that belong to the same clone than the leukemic monocytes seem to have immunosuppressive properties ressembling those of the myeloid-derived suppressor cells (MDCS) described in solid tumours. Whether these immature granulocytes contribute to autoimmune manifestations or immunoescape and progression of CMML is a conendrum and remains to be determined.

In this context, the proposed project aims at identifying news insights into the pathophysiology of CMML through a better definition of the phenotype and function of monocytes and immature granulocytes that characterize this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed or undergoing treatment in the Clinical Hematology department of the participating establishments

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic myelomonocytic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-11-05 (Actual); Primary Completion 2018-11-05 (Estimated); Study Completion 2018-11-05 (Estimated)

PRIMARY OUTCOMES:
Characterization of molecular mechanisms | at 3 years
  Characterization of the molecular mechanisms involved in the lack of differentiation of monocytes originating from patients with CML.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No